CLINICAL TRIAL: NCT03322956
Title: The Measurable Impact of a Protocoled Multimodal Physiotherapeutic Intervention on the Quality of Life in Patients With Non- Specific Chronic Low Back Pain. A Small RCT Study.
Brief Title: Effect of Physiotherapeutic Interventions on Quality of Life in Patients With Chronic Low Back Pain. (Study 1)
Acronym: CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Approved by the Committee of Medical Ethics University Hospital University of Brussels, B.U.N. 143201627110. (Unknown); Insurance on experiment on human subjects by ethias liability policy: 45.147.458 (Unknown); The EuroQol Research Foundation (Other); This research is supported by the Fysio Science Institute® and is a non-profit institution. (Unknown)
Responsible Party: Principal Investigator, Robbert van Amstel, Physical therapist, Master of science and manual therapist student, Vrije Universiteit Brussel
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EBP4MTOR01
Record Dates: First submitted 2017-10-07; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Physical Therapy; Chronic Low Back Pain; Quality of Life; Range of Motion; Pain Intensity
Keywords: Low back/lumbar spine; Multimodal Physical therapy; Quality of life; Range of Motion; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: One way, mixed, Randomized Controlled Trial(RCT), intention to threat design, level 2b.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (EGR) (Experimental): Physical therapy intervention.
  In the experimental group (EGR), the 4MTOR® treatment method will be used for LBP. This 4MTOR® uses the following steps in a decision tree: T1 Testing (Physiotherapeutic examination), T2 Triggering (Manual Techniques), T3 Taping (Elastic Tape) and T4 Training (medical rehabilitation exercises).
  Interventions: Other: Physioterapy intervention
- Sham group (SGR) (Sham Comparator): Physical therapy intervention.
  The participants in the SGR received a sham multimodal physiotherapeutic intervention as control intervention, in which Sham technique were applied. The interventions consisted of combining Sham manual interventions, elastic tapes according to Kaze and Evidence Based Practice Therapy. The protocol in the SGR follows the similar steps: Testing, Taping, Triggering and Training like the 4MTOR®.
  Interventions: Other: Physioterapy intervention

INTERVENTIONS:
Other: Physioterapy intervention — In the experimental group (EGR), the 4MTOR® treatment method will be used for LBP. This 4MTOR® uses the following steps in a decision tree: T1 Testing (Physiotherapeutic examination), T2 Triggering (Manual Techniques), T3 Taping (Elastic Tape) and T4 Training (medical rehabilitation exercises).
  The participants in the SGR received a sham multimodal physiotherapeutic intervention as control intervention, in which Sham technique were applied. The interventions consisted of combining Sham manual interventions, elastic tapes according to Kaze32 and Evidence Based Practice Therapy (Appendix III). The protocol in the SGR follows the similar steps: Testing, Taping, Triggering and Training like the 4MTOR®.

SUMMARY:
The purpose of this study is to investigate the effect on QoL, PI and the AROM° in patients with non-specific chronic low back pain. This after following an episode of 6 weeks 2 times a week physiotherapeutic back rehabilitation according to the 4 times T method by orthopedic disorder ® (4MTOR®). The results in this research will be analyzed and reported. In this study, 7 dependent variables will be independently examined relative to 2 independent variables.

DETAILED DESCRIPTION:
The purpose of this small RCT is to investigate whether this is a good research design and procedure to measure the effect on QoL, PI and the AROM° in patients with NSP-CLBP. This after following an episode of 6 weeks twice a week physiotherapeutic back rehabilitation according to the 4MTOR®. The results in this research will also be analysed and reported. The research design and procedure will be useful when this small RCT shows that the 4MTOR® can positively influence the QoL,PI and the AROM° with a p value <α = 0.05 in NSP-CLBP patients.

Primary variable is the QoL these are measured using the EQ-5D-3L which consists of the EQ-5D-index and the EQ visual analogue scale (EQ-VAS). The EQ-5D-3L questionnaire is developed by Euroqol Group. Secondary outcome measures are the AROM° of the active trunk flexion and trunk extension measured with a bubble inclinometer. Also, the PI will be scored by the patient during flexion and extension by means of the Verbal Pain Scale scaled 0-10 (VRS). The outcomes will be measured within 7 weeks in all participants. The measurements take place during week 0 the baseline measurement (W0), week 3 the intermediate measurement (W3) and finally week 7 the post measurement (W7). All participants were fully informed for the research and agreed by signing the "informed consent" (Appendix Ia). The research was approved by the Committee of Medical Ethics University Hospital University of Brussels, B.U.N. 143201627110.

Inclusion and exclusion criteria. Participants are included when they meet the following criteria: NSP-CLBP from 12 weeks and longer that are continuously present (with and without recurrent complaints), Age between 20 and 60 years and not yet treated by the 4MTOR®. Participants are excluded when they meet the following criteria: Radiological disturbing pain beyond knee, extremely serious neurological disorder symptoms, overall malaise, spinal cord malignancy, unexplained weight loss, prolonged corticosteroid use, osteoporotic vertebral fracture, spondylitis ankylopoetics, spinal stenosis, rheumatic arthritis, vertebral fracture and severe deformity of the spinal cord.

Recruitment. Patients recruitment: The subjects are recruited from orthopedic hospitals departments in Utrecht the Netherlands. Participants will be asked if they want to refer NSP-CLBP patients for this research and by advertisement in an Dutch-language newspaper (Appendix II). Also, NSP-CLBP patients who applied for physical therapy were asked if they wanted to participate in this research. A call form has been prepared for this purpose (Appendix III). All subjects were asked if they would like to participate in this research. The subjects has been authorized to perform medical physiotherapeutic treatment. This has been done by signing a statement of agreement, as previously stated. Personal data will not be included in this research and are protected by researchers and the Committee of Medical Ethics University Hospital University of Brussels.

Therapist recruitment Experimental intervention group: This physiotherapist has been educated and qualified in the KNGF accredited multimodal intervention according to the 4MTOR®. The physiotherapist has at least 2 years of work experience with the use of the 4MTOR® decision tree.

Therapist recruitment SHAM intervention group: This is Health Care registered physiotherapist and has at least 3 years work experience and is familiar with the KNGF Low Back pain, 2013 guidelines (KNGF_LBP)74. Both therapists were informed about their work protocol and have agreed to the implementation of the interventions by signing an informed consent.

In the experimental group (EGR), the 4MTOR® treatment method will be used for LBP. This 4MTOR® uses the following steps in a decision tree: T1 Testing (Physiotherapeutic examination), T2 Triggering (Manual Techniques), T3 Taping (Elastic Tape) and T4 Training (medical rehabilitation exercises).

The participants in the Sham group (SGR) received a sham multimodal physiotherapeutic intervention as control intervention, in which Sham technique were applied. The interventions consisted of combining Sham manual interventions, elastic tapes according to Kaze32 and Evidence Based Practice Therapy (Appendix III). The protocol in the SGR follows the similar steps: Testing, Taping, Triggering and Training like the 4MTOR®.

Primary:

- EQ 5d-5L questionnaire

Secondary:

Thoracolumbo-pelvic flexion, inclinometry Thoracolumbo-pelvic extension, inclinometry Isolated lumbar flexion, inclinometry Verbal pain score flexion, VRS 0-10 Verbal pain score extension, VRS 0-10

Research design. This research is a one way, Mixed, real experimental design One way design (Independent Groups variables). Mixed Design: Baseline Week 0 - Week 3 - Week 7 Within groups: difference in time Between groups: difference between groups.

The RMANOVA-MD power analysis was performed using the following values: Power.81, Alpha 0.50, Sample size effect f2 =.25, resulting in a minimum of 28 participants, Fcritical = 3.175 and an actual power of .82 . Cohen advises a medium-sized effect size (f2 = .25) in a RMANOVA-MD. 10% will be added to these 28 participants (n = 30), towards the possible dropouts. The NSP-CLBP participants are divided into 2 groups.

ELIGIBILITY:
Inclusion Criteria:

Participants are included when they meet the following criteria:

* NSP-CLBP from 12 weeks and longer that are continuously present (with and without recurrent complaints)
* Age between 20 and 60 years
* Not yet treated by the 4MTOR®.

Exclusion Criteria:

Participants are excluded when they meet the following criteria:

* Radiological disturbing pain beyond knee
* Extremely serious neurological disorder symptoms
* Overall malaise
* Spinal cord malignancy
* Unexplained weight loss
* Prolonged corticosteroid use
* Osteoporotic vertebral fracture
* Spondylitis ankylopoetics
* Spinal stenosis
* Rheumatic arthritis
* Vertebral fracture
* Severe deformity of the spinal cord

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
First measurment: Quality of life, EQ-5D-3L-index | Timespad registration: Week 0/baseline measurement (W0) - week 3/intermediate measurement (W3)
  The EQ-5D-3L-index will analyze the participants Quality of life (QoL). Each question in the EQ-5D-3L-index includes one dimension of QoL: mobility, self-care, daily activities, pain/discomfort & anxiety/depression. Each dimension has 3 levels ( having no problems, having some or moderate problems, being unable to do/having extreme problems) and gets a separate score.The scores can be combined in combination with an assessment of the health status they represent, this rating is expressed in weight or utility (1,000 = no problems at all) to (-0,329= extreme problems). Description of the QoL can be transformed into a QoL assessment by means of a formula. These ratings are based on judgments of the general population of all possible combinations of QoL on the different dimensions. An improvement in quality of life will be assumed when p<α=0.05.
  Within time: W0-W3 Between groups: EGR versus SGR. The results are shown for all variables in a table.
Second measurment: Quality of life, EQ-5D-3L-index | Timespad registration: Week 3/intermediate measurement (W3) - Week 7 post measurment
  The EQ-5D-3L-index will analyze the participants Quality of life (QoL). Each question in the EQ-5D-3L-index includes one dimension of QoL: mobility, self-care, daily activities, pain/discomfort & anxiety/depression. Each dimension has 3 levels ( having no problems, having some or moderate problems, being unable to do/having extreme problems) and gets a separate score.The scores can be combined in combination with an assessment of the health status they represent, this rating is expressed in weight or utility (1,000 = no problems at all) to (-0,329= extreme problems). Description of the QoL can be transformed into a QoL assessment by means of a formula. These ratings are based on judgments of the general population of all possible combinations of QoL on the different dimensions. An improvement in quality of life will be assumed when p<α=0.05..
  Within time: W3-W7 Between groups: EGR versus SGR. The results are shown for all variables in a table.
Third measurment: Quality of life, EQ-5D-3L-index | Timespad registration: Week 0/baseline measurement (W0)- Week 7 post measurment
  The EQ-5D-3L-index will analyze the participants Quality of life (QoL). Each question in the EQ-5D-3L-index includes one dimension of QoL: mobility, self-care, daily activities, pain/discomfort & anxiety/depression. Each dimension has 3 levels ( having no problems, having some or moderate problems, being unable to do/having extreme problems) and gets a separate score.The scores can be combined in combination with an assessment of the health status they represent, this rating is expressed in weight or utility (1,000 = no problems at all) to (-0,329= extreme problems). Description of the QoL can be transformed into a QoL assessment by means of a formula. These ratings are based on judgments of the general population of all possible combinations of QoL on the different dimensions. An improvement in quality of life will be assumed when p<α=0.05.
  Within time: W3-W7 Between groups: EGR versus SGR. The results are shown for all variables in a table.
First measurment: EQ- visual analogue scale (VAS) | Timespad registration: Week 0/baseline measurement (W0) - week 3/intermediate measurement (W3)
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical (0-100 score), visual analogue scale with endpoints labelled 'the best health (100) you can imagine' and 'the worst health you can imagine (0) '. This information can be used as a quantitative measure of health as judged by the individual respondents. An improvement in quality of life will be assumed when p<α=0.05. For the EQ-VAS we used the minimum important change (MIC) for VAS 15 points
  Within time: W0-W3 Between groups: EGR versus SGR. The results are shown for all variables in a table.
Second measurment: EQ- visual analogue scale (VAS) | Timespad registration: Week 3/intermediate measurement (W3) - Week 7 post measurment
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical (0-100 score), visual analogue scale with endpoints labelled 'the best health (100) you can imagine' and 'the worst health you can imagine (0) '. This information can be used as a quantitative measure of health as judged by the individual respondents. An improvement in quality of life will be assumed when p<α=0.05. For the EQ-VAS we used the minimum important change (MIC) for VAS 15 points
  Within time: W3-W7 Between groups: EGR versus SGR. The results are shown for all variables in a table.
Third measurment: EQ- visual analogue scale (VAS) | Timespad registration: Week 0/baseline measurement (W0)- Week 7 post measurment
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical (0-100score), visual analogue scale with endpoints labelled 'the best health (100) you can imagine' and 'the worst health you can imagine (0) '. This information can be used as a quantitative measure of health as judged by the individual respondents. An improvement in quality of life will be assumed when p<α=0.05. For the EQ-VAS we used the minimum important change (MIC) for VAS 15 points
  Within time: W0-W7 Between groups: EGR versus SGR. The results are shown for all variables in a table.

SECONDARY OUTCOMES:
AROM° thoracolumbar-pelvic flexion (TLPF) | Timespad registration: Week 0/baseline measurement (W0), week 3/intermediate measurement (W3) and week 7/ post measurement (W7).
  AROM° Thoracolumbar-pelvic flexion. The inclinometer placed on L1 / T12 with the tape between the inclinometer arcus and was set to 0°. During the test, the investigator kept the inclinometer on L1 / T12 while instructing the subject to bend forward with the arms in hanging position.
  The changes in our variables will be analyzed within time and between groups.
  Within time: W0-W3, W0-W7 and W3-W7, Between groups: EGR versus SGR. The results are shown for all variables in a table. The analysis for all variables is significant when p<α=0.05.
AROM° thoracolumbar- pelvic extension (TLPE) | Timespad registration: Week 0/baseline measurement (W0), week 3/intermediate measurement (W3) and week 7/ post measurement (W7).
  AROM° Thoracolumbar-pelvic extension. The inclinometer placed on L1 / T12 with the tape between the inclinometer arcus and was set to 0 °. During the test, the investigator kept the inclinometer on L1 / T12 while instructing the subject to put his hands on his pelvis and bend backward.
  The changes in our variables will be analyzed within time and between groups. Within time: W0-W3, W0-W7 and W3-W7, Between groups: EGR versus SGR. The results are shown for all variables in a table. The analysis for all variables is significant when p<α=0.05.
AROM° isolated lumbar flexion(ILF) | Timespad registration: Week 0/baseline measurement (W0), week 3/intermediate measurement (W3) and week 7/ post measurement (W7).
  AROM° Isolated lumbar flexion test. The inclinometer was moved to labeled S1 / S2 and the inclinometer was set to 0 °. During the test, the investigator held the inclinometer on S1 / S2 while instructing the subject to bend forward. The formula ∑▒〖T12/L1〗 - S1/S2 was used.
  The changes in our variables will be analyzed within time and between groups. Within time: W0-W3, W0-W7 and W3-W7, Between groups: EGR versus SGR. The results are shown for all variables in a table. The analysis for all variables is significant when p<α=0.05.
Pain intensity extension (0-10) | Timespad registration: Week 0/baseline measurement (W0), week 3/intermediate measurement (W3) and week 7/ post measurement (W7).
  Before the participant gave a PI number to the active extension, the Verbale pain Rating Scale (VRS) scale was shown. Thereafter the movement was performed as described in the protocol. After completing the active extension, the participant gave a VRS score regarding the PI. Studies have shown that a score of 0-10 must be at least 30% reduction with a range between 1 to 4.5 on a maximum of 10 points12. In this study, we used the Minimal Important Change (MIC) of 2 points (4.5 <) were chosen. .
  The changes in our variables will be analyzed within time and between groups.
  Within time: W0-W3, W0-W7 and W3-W7, Between groups: EGR versus SGR. The results are shown for all variables in a table. The analysis for all variables is significant when p<α=0.05.
Pain intensity flexion (0-10) | Timespad registration: Week 0/baseline measurement (W0), week 3/intermediate measurement (W3) and week 7/ post measurement (W7).
  Before the participant gave a PI number to the active flexion , the Verbale pain Rating Scale (VRS) scale was shown. Thereafter the movement was performed as described in the protocol. After completing the active flexion, the participant gave a VRS score regarding the PI. Studies have shown that a score of 0-10 must be at least 30% reduction with a range between 1 to 4.5 on a maximum of 10 points12. In this study, we used the Minimal Important Change (MIC) of 2 points (4.5 <) were chosen. .
  The changes in our variables will be analyzed within time and between groups.
  Within time: W0-W3, W0-W7 and W3-W7, Between groups: EGR versus SGR. The results are shown for all variables in a table. The analysis for all variables is significant when p<α=0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P. Vaes, PhD, Study Director — University of Brussels, faculty of Rehabilitation science and physical therapy, faculty of Pharmacy and medicine, Brussels, Belgium
Locations (1):
- Peter Vaes, Jette, Brussels Capital, Belgium